CLINICAL TRIAL: NCT01710956
Title: Randomized Phase II Study of Once Daily Accelerated Fractionation With Concomitant Boost to the Gross Tumor Volume Compared With Twice Daily Hyperfractionation in Concurrent Chemoradiation in Patients With Limited Disease Small Cell Lung Cancer
Brief Title: Once Daily Accelerated Fractionation With Concomitant Boost to the Gross Tumor Volume Compared With Twice Daily Hyperfractionation in Concurrent Chemoradiation in Patients With Limited Disease Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Kwan Ho Cho, PI, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-11-531
Record Dates: First submitted 2012-10-16; First posted 2012-10-19 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Limited Disease Small Cell Lung Cancer
Keywords: concurrent chemoradiation in patients with limited disease small cell lung cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1(with twice-daily TRT) (Experimental)
  Interventions: Radiation: Arm 1: with twice-daily thoracic radiotherapy/ Arm 2: with once-daily thoracic radiotherapy
- Arm 2 (with once-daily TRT) (Experimental)
  Interventions: Radiation: Arm 1: with twice-daily thoracic radiotherapy/ Arm 2: with once-daily thoracic radiotherapy

INTERVENTIONS:
Radiation: Arm 1: with twice-daily thoracic radiotherapy/ Arm 2: with once-daily thoracic radiotherapy — Arm 1: with twice-daily thoracic radiotherapy daily 1.5gy/fr. bid, total 45gy(30fr during 3weeks) Arm 2: with once-daily thoracic radiotherapy daily 2.4gy/fr. qd, total 60gy(25fr during 5weeks)

SUMMARY:
Non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically (if cannot be proven histologically, at least twice positive findings on fine needle aspiration or sputum cytology) confirmed SCLC
* Limited stage (Clinical stage I-IIIb, lesion limited to one side of thorax, e.g. Excluding T4 disease with malignant pleural effusion or N3 disease with contralateral hilum/supraclavicular lymph node invasion).
* Measurable or assessable lesion
* Age over 18 years old
* Performance status (ECOG scale): 0~2
* Adequate organ functions: ANC ≥ 1500/ul, PLT ≥ 100 x 103/u, Total Bilirubin ≤ 1.5 mg/dl, Creatinine ≤ 1.5 mg/dl
* Inclusion of tumor within the limited radiation field without significant loss of pulmonary function (confirmed by radiation oncologist)
* Sexually active fertile men and women using a contraceptive method
* Patients should sign a written informed consest before study entry

Exclusion Criteria:

* T4 disease with malignant pleural effusion; N3 disease with contralateral hilum/supraclavicular lymph node invasion
* Lesion with mixed small cell nonsmall cell feature (pathologically)
* prior chemotherapy or radiation therapy.
* Pericardial or pleural effusion on chest X-ray image regardless of cytological finding
* T4 disease with tumor invasion to great vessels, heart, trachea, or esophagus; Concerns about possible perforation by tumor necrosis
* Severe comorbidities such as cardiac disease with symptom, myocardiac infarction within 6 months, chronic obstructive pulmonary disease with FEV1 less than 1.0ℓ, or uncontrolled bronchospasm of unaffected lung
* With atelectasis that makes GTV unidentifiable
* Other primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 3 years ago without recurrence)
* Uncontrolled psychiatric disorder, serious head injury, chronic alcoholism, drug addiction and central nervous system disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 5years after chemoradiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Kwan Ho Cho, M.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Canter, Korea, Ilsan-ro 323, Ilsandoung-gu, Goyang-si, Gyeonggi-do, South Korea